CLINICAL TRIAL: NCT02726035
Title: Evaluation of Naltrexone as a Treatment for Self-Injurious Behavior
Acronym: NTX-SIB
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI deceased
Sponsor: Western Michigan University School of Medicine (Other)
Collaborators: Kalamazoo Community Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BorgessIRB-2014-0672
Record Dates: First submitted 2016-03-18; First posted 2016-04-01 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Self-injurious Behavior; Self Mutilation
Keywords: Self-injurious behavior; Self mutilation; naltrexone
MeSH Terms: conditions — Self-Injurious Behavior; Self Mutilation | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 A-ABAB (Experimental): After 4 week open label oral naltrexone run-in, participants are randomized to 2 groups (50% each). Group 1 will receive oral naltrexone 50 mg daily during weeks 5-7 (3 weeks). They will switch to placebo for weeks 8-10, then return to naltrexone for weeks 11-13, then placebo for weeks 14-16 (i.e., A-ABAB double crossover design, participants act as own controls). Study drug and placebo will be encapsulated so as to appear identical.
  Interventions: Drug: Naltrexone; Other: Placebo
- Group 2 A-BABA (Experimental): After 4 week open label oral naltrexone run-in, participants are randomized to 2 groups (50% each). Group 2 will receive oral placebo once daily during weeks 5-7. They will then be switched to oral naltrexone 50 mg daily for weeks 8-10, then return to placebo for weeks 11-13, then naltrexone for weeks 14-16 (i.e., A-BABA double crossover design, participants act as own controls). Study drug and placebo will be encapsulated so as to appear identical.
  Interventions: Drug: Naltrexone; Other: Placebo

INTERVENTIONS:
Drug: Naltrexone — oral naltrexone 50 mg daily
  Other Names: Revia
Other: Placebo — oral placebo (appearing identical to naltrexone) once daily

SUMMARY:
The proposed study examines the effect of oral naltrexone on self-injurious behavior (SIB) in adolescents and adults of normal intelligence.

DETAILED DESCRIPTION:
The proposed study examines the effect of oral naltrexone on self-injurious behavior (SIB) in adolescents and adults of normal intelligence. It is designed as a pilot study and will provide preliminary data for a larger scale clinical trial if found to be effective in the pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Thirteen years of age or older
* Actively engaged in SIB at a rate of, on average, at least two events per week for at least 3 months
* Has internet access in a secure and private manner
* Lives within a reasonable distance from Kalamazoo (to make the five clinic visits convenient) and plans to remain in the area throughout the next 4-5 months

Exclusion Criteria:

* Under the age of 13
* Currently pregnant (confirmed with initial urine pregnancy test), lactating, or planning to become pregnant in the next 4 months
* Active hepatitis or liver disease
* Prior history of recently active opioid dependence
* Current prescription, non-prescription, or illicit opioid use, (i.e., acute use within the past 14 days or chronic use within the last 30 days), including all opioid analgesics, certain cough and cold remedies (e.g., codeine), and certain anti-diarrheal preparations (e.g., loperamide). Currently taking an opioid antagonist for alcohol or opioid dependence or having taken one in the last 14 days
* Current use of leflunomide (Arava), droperidol (Droleptan), diazepam (Valium), thioridazine (Mellaril, Novoridazine, Thioril) (26)
* Any report of clinically significant medical condition or medication regimen which might cause undue risk or affect ability to participate in this clinical trial
* On initial laboratory examination, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels more than one standard deviation (SD) above the upper limit of normal
* Unable to meet a 22-week requirement to log journal entries daily, to be available by phone a minimum of once weekly during the first month, and to be present at clinical sites once every three weeks for 12 weeks, for a total of 5 visits
* Infrequent SIB, lack of secure Internet access, or living a significant distance from the Kalamazoo area (does not meet inclusion criteria)
* Unwilling or parent/guardian unwilling to participate in research requirements.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02-22 (Actual); Primary Completion 2015-06-30 (Estimated); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Comparison of self-injury rates by condition | For each 3 week trial, average rates calculated over weeks 2-3 only (14 day period).
  naltrexone rate vs. placebo rate

SECONDARY OUTCOMES:
Comparison of self-injury rates by trial within condition | Average rates calculated for weeks 2-3 of each 3 week trial (14 day period)
  1st naltrexone trial vs. 2nd & 1st placebo trial vs. 2nd

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Liepman, MD, Principal Investigator — Western Michigan University School of Medicine; Chris A. Karampahtsis, MD, MPH, Principal Investigator — Western Michigan University School of Medicine
Locations (1):
- Borgess Research Institute, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No